CLINICAL TRIAL: NCT07043660
Title: Promoting Adoptive Parents' Well-being: A Randomized Controlled Pilot Trial to Evaluate a Mindful Parenting Post-adoption Intervention
Brief Title: Preliminary Efficacy of AdoptMindful2Care: A Mindful Parenting Post-adoption Intervention for Adoptive Parents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Bárbara Caetano, Principal Investigator, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pAdoptMindful2Care/154436/2022; UI/BD/154436/2022 (Other Grant/Funding Number: Fundação para a Ciência e a Tecnologia); CEECIND/02463/2017 (Other Grant/Funding Number: Fundação para a Ciência e a Tecnologia)
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Parenting Stress
Keywords: parenting stress; mindful parenting intervention; adoptive parents; postadoption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AdoptMindful2Care Intervention (Experimental): Adoptive mothers and fathers will receive a structured 8-week group program based on mindful parenting principles, delivered in person during the study period
  Interventions: Behavioral: AdoptMindful2Care
- Waiting list group (Other): Adoptive mothers and fathers will not receive the intervention during the study period but will be offered and receive AdoptMindful2Care after the final follow-up assessment is completed.
  Interventions: Behavioral: AdoptMindful2Care

INTERVENTIONS:
Behavioral: AdoptMindful2Care — AdoptMindful2Care is a mindful parenting post-adoption intervention with eight weekly group sessions (approximately 90 minutes each), delivered in person by trained psychologists, plus one follow-up session held two months after completion. The intervention integrates psychoeducation, mindfulness-based exercises, mindful parenting and self-compassion practices, as well as strategies informed by Cognitive Behavioral Therapy (CBT). The program is designed to help adoptive parents reduce parenting stress and promote positive parenting practices.

SUMMARY:
Adoptive parents often face additional challenges related to the adoption process, which can increase their vulnerability to parenting stress and negatively affect their parenting practices and overall family well-being. These risks highlight the urgent need to implement post-adoption interventions that reduce parenting stress and promote both parental well-being and positive parenting practices.

In this study, the research team aims to evaluate the preliminary efficacy of AdoptMindful2Care, a new 8-week, face-to-face, group-based psychological intervention grounded in the principles of mindful parenting. This pilot randomized controlled trial, which uses a two-arm design, serves as a preliminary step before conducting the full-scale RCT planned for AdoptMindful2Care.

The investigators will invite both mothers and fathers to participate if they have at least one adoptive child between the ages of 2 and 17 and if the legal adoption decree was finalized in court at least 12 months before enrollment. The investigators will target parents who report moderate to high levels of parenting stress. With the support of all Portuguese governmental adoption agencies, the researchers plan to recruit a minimum of 78 families.

After parents express interest in participating, the investigators will screen them to assess their levels of parenting stress. For those who meet the initial criteria, the investigators will conduct a structured clinical interview (SCID-5-CV) to rule out severe mental illness. If participants meet all inclusion criteria and present no exclusion criteria, the investigators will proceed with a final interview to guide them through the informed consent process.

The investigators will randomly assign eligible participants to either the intervention group (AdoptMindful2Care) or a waitlist control group (who will receive the intervention after the study concludes). All participants will be informed that they will be randomized to one of the study groups and that they will only be included if they give informed consent to participate in the study. The investigators will deliver the intervention in person, in a group format, through eight weekly sessions and one follow-up session, each lasting approximately 90 minutes.

All participants will complete assessments at three time points: baseline, post-intervention, and 2-month follow-up. These assessments will include self-report measures (e.g., parenting stress) and hetero-report measures (e.g., children's emotional and developmental difficulties).

ELIGIBILITY:
Inclusion Criteria:

* Being a mother and/or father of at least one adoptive child aged between 2 and 17 years old, inclusive.
* The adoption must have been legally finalized in court for more than 12 months.
* Presence of moderate to high levels of parenting stress.

Exclusion Criteria:

* Presence of a severe mental disorder (e.g., schizophrenia, substance abuse, bipolar disorder).
* Are receiving another psychological intervention focused on parenting issues.
* Are receiving technical support under a child and youth protection measure that involves the institutionalization of the child/youth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in parenting stress | Baseline, 2 and 4 months
  Measured with Parenting Stress Index - Short Form. The 36 PSI-SF items are divided into three subscales: parenting difficulties, dysfunctional parent-child interactions, and child difficulties. Items are rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree), with higher total scores indicating higher levels of parenting stress.

SECONDARY OUTCOMES:
Changes from baseline in mindful parenting | Baseline, 2 and 4 months
  Measured with Interpersonal Mindfulness in Parenting Scale (IMP). The IMP is a 31-item self-report questionnaire; each item is rated on a 5-point Likert scale ranging from 1 (never true) to 5 (always true), with a higher total score indicating higher levels of mindful parenting.
Changes from baseline in anxiety and depressive symptoms | Baseline, 2 and 4 months
  Measured with Hospital Anxiety and Depression Scale (HADS). HADS is a 14-item self-report questionnaire comprising 2 subscales: anxiety and depression. Each subscale consists of 7 items rated on a 4-point Likert scale. Subscale scores are calculated separately, with higher scores indicating higher levels of anxiety or depressive symptoms, respectively.
Changes from baseline in coparenting | Baseline, 2 and 4 months
  Measured with Questionnaire on Parental Perceptions of Coparenting (QPPC). QPPC is a 14-item self-report questionnaire; each item is rated on a 5-point Likert scale ranging from 1 (never) to 5 (always), with a higher total score indicating greater perceived quality of coparenting.
Changes from baseline in children's emotional and behavioral difficulties | Baseline, 2 and 4 months
  Measured with Strengths and Difficulties Questionnaire (SDQ). SDQ is a 25-items self-report questionnaire available in two versions (for ages 2-4 and 4-17), which share the same structure, scoring method, and interpretation. The SDQ comprises five subscales: Emotional Symptoms, Conduct Problems, Hyperactivity/Inattention, Peer Relationship Problems, and Prosocial Behavior. Items are rated on a 3-point Likert scale, from 0 (Not true) to 2 (Very true). The total difficulties score is calculated by summing the scores from all subscales except Prosocial Behavior, with higher scores indicating greater emotional and behavioral difficulties.
Changes from baseline in self-compassion | Baseline, 2 and 4 months
  Measured with the Self-Compassion Scale - Short Form (SCS-SF). SCS-SF is a 12-item self-report questionnaire organized into six subscales: self-kindness, self-judgment, mindfulness, isolation, and overidentification. Items are rated on a 5-point Likert scale ranging from 1 (Almost never) to 5 (Almost always), with higher total scores indicating greater levels of self-compassion.
Changes from baseline in emotional regulation | Baseline, 2 and 4 months
  Measured with the Difficulties in Emotion Regulation Scale - Short Form (DERS-SF). DERS-SF is an 18-item self-report questionnaire; each item is rated on a 5-point Likert scale ranging from 1 (Almost never) to 5 (Almost always), and a higher total score is indicative of more difficulties in emotion regulation.
Changes from baseline in mindfulness | Baseline, 2 and 4 months
  Measured with the Mindful Attention and Awareness Scale (MAAS). MAAS is a 15-item self-report questionnaire; each item is rated on a 6-point Likert scale ranging from 1 (almost always) to 6 (almost never), with a higher total score indicating greater levels of mindfulness.
Acceptability of the intervention | 2 months
  Measured through specific questions (developed by the researchers) to assess acceptability.

CONTACTS AND LOCATIONS:
Locations (4):
- Portugal (4):
  - Instituto da Segurança Social - Centro Distrital de Aveiro, Aveiro
  - Faculty of Psychology and Education Sciences, University of Coimbra, Coimbra
  - Instituto da Segurança Social, I.P., Lisbon
  - Instituto da Segurança Social - Centro Distrital do Porto, Porto

IPD SHARING:
Plan to Share IPD: Undecided
After the conclusion of the trial, the investigators plan to share the results of the study both with scientific community and health professionals.